CLINICAL TRIAL: NCT05714215
Title: Italian Translation and Transcultural Validation of the Simplified Evaluation of Consciousness Disorders (SECONDs) Scale: a Multicentre Study
Brief Title: SECONDs' Italian Translation and Transcultural Validation
Acronym: IT-SECONDs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Carlo Besta Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IT-SECONDs
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Disorder of Consciousness
Keywords: Disorders of Consciousness; Scale; Validation; diagnosis
MeSH Terms: conditions — Consciousness Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The coma recovery scale-revised (CRS-R) is the recommended diagnostic scale for consciousness but it requires time, training, and provides total scores that do not always reflect the correct level of consciousness. Recently, a new short-term assessment tool for consciousness assessment has been validated, which could easily be implemented in daily practice to determine the level of consciousness in severely brain injured individuals: the simplified evaluation of consciousness disorders (SECONDs) .Its administration should be significantly shorter than CRS-R and accurate to allow monitoring of consciousness in the subacute / chronic phase. The SECONDs scale was constructed by selecting the items that, based on the latest scientific evidence, are most frequently associated with a minimally consciousness state. In fact, recent studies have shown that 5 items of the CRS-R allow to identify 99% of individuals with minimally consciousness state 1) reproducible movement on command, 2) visual pursuit 3) visual fixation 4) automatic motor response, and 5) localization to pain) 12. In addition, some changes have been introduced such as 1) the assessment of fixation and visual tracking through the use of the mirror 2) the use of autobiographical questions for the assessment of communication 3) the reduction of the number of orders on command to 2 of 3 instead of 3 out of 4 as in the CRS-R. All these changes have been made to minimize time for administration without compromising the accuracy of consciousness detection, to improve feasibility in clinical practice, and also to limit fatigue, which could produce better patient concentration and collaboration.

The aim of the multicentre study is to carry out a cross-cultural translation of the SECONDs assessment scale into Italian and to perform a validation between operators of different professions of the Italian version. validation will be conducted on a group of patients with prolunged disorders of consciousness in the subacute phase admitted to two units of severe acquired brain injuries of the don Carlo Gnocchi Foundation of Florence and Sant'Angelo dei Lombardi, and in the chronic phase IRCCS foundation Carlo Besta neurological institute

DETAILED DESCRIPTION:
The first phase involves the Italian translation of the SECONDs scale through a rigorous multi-stage review and the drafting of the working and final versions. First, the original scale will undergo a forward translation into Italian by a certified translator. The Italian version obtained will then be discussed by the team of experts from the 3 centers participating in the study for transcultural adaptation. Then the revised Italian version will be subsequently back translated into the original language by another certified translator blinded from the original version. Any discrepancy will be thoroughly discussed between the interdisciplinary Italian group and with the external expert from the group that originally developed the scale, and the Italian version shall be re-defined, with the aim of determining the conceptual, semantic, and operational equivalence of the translated scale. (Phase 1) The second phase involves a pilot study in which the final Italian version of the identified scale will be administered to a small group of patients to determine its intra and interoperative validity (Phase 2A) Subsequently, the multicentre validation of the Italian scale is envisaged on a larger group of patients, 38 admitted to inpatient intensive rehabilitation in the subacute phase (don Gnocchi foundation) and 22 admitted to outpatient rehabilitation in the chronic phase (Istituto Besta) (Phase 2B).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe acquired brain injury
* Diagnosis of a disorder of consciousness

  •> 28 days from the acute event
* age> 18 years
* No history of neurological or psychiatric deficits
* Mother tongue: Italian
* Clinical stability (eg, absence of mechanical ventilation, sedation, infection, ensuing seizures).
* Signature of the informed consent by the legal representative

Exclusion Criteria:

• Appearance of a second brain event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the pilot intra and inter-rater validation study (Phase 2A), the enrollment of 10 consecutive patients (5 Florence, 2 Sant'Angelo and 3 Besta) is envisaged, subject to the signature of the informed consent of the legal representative.
  For the second phase of multicentre validation, the recruitment of 60 consecutive or distributed patients is foreseen, Florence: 28; Sant'Angelo: 10 and Istituto Besta: 22.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The concurrent validity of the transcultural adaptation of the SECONDs scale with the CRS-R (correlation coefficient for Spearman's ranks) | 21 months
  The endpoint of the study is the creation of a valid and reliable transcultural adaptation of the SECONDs scale
the indexes of agreement between inter and intra examiners (index K) | 21 months
  The endpoint of the study is the creation of a valid and reliable transcultural adaptation of the SECONDs scale

CONTACTS AND LOCATIONS:
Overall Officials: Bahia Hakiki, Dr, Principal Investigator — IRCCS-Fondazione Don Gnocchi-Florence; Bahia Hakiki, Dr, Study Director — IRCCS-Fondazione Don Gnocchi-Florence
Locations (1):
- IRCCS-don Gnocchi Foundation, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aubinet C, Cassol H, Bodart O, Sanz LRD, Wannez S, Martial C, Thibaut A, Martens G, Carriere M, Gosseries O, Laureys S, Chatelle C. Simplified evaluation of CONsciousness disorders (SECONDs) in individuals with severe brain injury: A validation study. Ann Phys Rehabil Med. 2021 Sep;64(5):101432. doi: 10.1016/j.rehab.2020.09.001. Epub 2021 Jul 28. PMID 32992025
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342